CLINICAL TRIAL: NCT06261632
Title: Safety and Efficacy of a Physiotherapy Intervention Through Blood Flow Restriction in Improving Muscle Strength in Patients With Hemophilic Knee Arthropathy: Multicenter Randomized Clinical Study
Brief Title: Blood Flow Restriction in Improving Muscle Strength of Patients With Hemophilic Knee Arthropathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hemo-Blood
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia
Keywords: Hemophilic arthropathy; Blood flow restriction; Physiotherapy; Muscular strength; Muscle activation; Range of Motion; Chronic pain; Functionality; Quality of life
MeSH Terms: conditions — Hemophilia A; Chronic Pain | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention will consist of carrying out a physiotherapy protocol, consisting of strength training through blood flow restriction, with an occlusion pressure of 40-50% of the LOP (Limb Occlusion Pressure) and a load of 20-30%. of 1RM performed ad hoc for patients with hemophilic arthropathy.
  The intervention protocol will be carried out in person under the supervision of the main researcher. The intervention will last 4 weeks, with a frequency of 3 weekly sessions. In total there will be 12 sessions lasting approximately 30-45 minutes
  Interventions: Other: Blood flow restriction
- Control group (No Intervention): The patients included in the control group will not receive any Physiotherapy intervention and will continue with their usual routine, being evaluated in the same periods as the rest of the patients.

INTERVENTIONS:
Other: Blood flow restriction — The intervention protocol through blood flow restriction in patients with hemophilic arthropathy will include performing squats and knee extension for 5-10 and 10 minutes respectively. In both exercises, 4 series will be performed (30, 15, 15, 15 repetitions) with 30 seconds of rest between series
  Arms: Experimental group

SUMMARY:
Background. The main physical sequela of patients with hemophilia is the development of a progressive, degenerative intra-articular lesion, known as hemophilic arthropathy). This sequela is manifested by chronic pain, limited range of motion, axial abnormalities, and periarticular muscle atrophy.

Objective. To assess the safety and effectiveness of an intervention through blood flow restriction, regarding the frequency of bleeding and the improvement in muscle activation and strength, range of motion, functionality, joint pain, joint status and the perception of quality of life in patients with hemophilic arthropathy. knee and ankle.

Study design. Randomized, multicenter, single-blind clinical study. Method. 60 patients with hemophilia A and B will be recruited in this study. Patients will be recruited in 6 regions of Spain. The dependent variables will be: bleeding frequency (self-registration), pain (measured with the visual analog scale and pressure algometer), quality of life (SF-36 scale), joint status (Hemophilia Joint Health Score scale), strength (dynamometer) and muscle activation (surface electromyograph), range of motion (goniometer) and functionality (Timed up and go test). Three evaluations will be carried out: pre-treatment, post-treatment and after a follow-up period of 4 weeks.

Expected results. Observe the safety of blood flow restriction in hemophilia patients. To analyze the efficacy of blood flow restriction in improving muscle strength and activation, range of motion, chronic pain, functionality, and the perception of quality of life in patients with hemophilic knee and ankle arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* People with a medical diagnosis of hemophilic knee arthropathy
* Adults (> 18 years)
* In prophylactic treatment regimen or on demand with FVIII/FIX concentrates.
* Failure to sign the informed consent document

Exclusion Criteria:

* Patients with neurological or cognitive alterations that prevent understanding of the questionnaires
* Amputee patients, epileptics or patients with severe vision problems
* Patients who are receiving physiotherapy treatment at the time of the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline hemarthrosis after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  self-registration will be used to evaluate the frequency of bleeding, and thus the safety of the technique. This self-registration will be given to each patient at the beginning of the study and they must fill in the number of hemarthrosis and their main characteristics: date, origin (traumatic or spontaneous) and location (knee or ankle). The self-registration will be delivered to the evaluator in each of the study evaluations (post-treatment and follow-up).

SECONDARY OUTCOMES:
Change from baseline pressure pain threshold after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With a pressure algometer (model Wagner FPN100) we will measure the pressure pain threshold, at the joint level and at a distance (in another part of the body). This device measures in Newton / cm2 the pressure at which the subject perceives pain under pressure. A pressure will be made on the chosen point, which we will increase at an approximate speed of 50kPa / s until the patient warns us that the sensation begins to be painful. Hemophilic arthropathy will be assessed in the knee (inner edge of the patella) and ankle (lateral malleolus).
Change from baseline muscle strength after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With a pressure dynamometer (microFET®2 Digital Handheld model) we will measure the strength of the quadriceps and triceps surae. This device measures in Newton the force that the patient exerts in the requested muscular action. The higher the value, the greater the muscle strength. We will carry out the measurements bilaterally. The patient will be asked 4 maximum isometric contractions of 5 seconds, with a rest of 30 seconds between them, against the dynamometer located in the hand of the evaluator
Change from baseline electrical activity of the muscles after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  Using surface electromyography (model SHIMMMER2, Shimmer, Ireland), we will evaluate the electrical activity of the musculature and its level of activation. The placement of the electrodes will be marked on the standing subjects, and they will be placed following the European recommendations for the use of the SEMG. A bipolar SEMG system will be used with circular electrodes 10 mm in diameter, 20 mm apart, placed longitudinally, in the direction of the fibers of the studied muscle, and with a remote reference electrode
Change from baseline range of motion after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  The range of motion of the knee joint will be measured using a universal goniometer, using the protocol for measuring joint motion described by the American Academy of Orthopaedic Surgeons
Change from baseline joint status after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With the Hemophilia Joint Health Score scale, specific for its use in patients with hemophilia, the joint status of patients with hemophilic arthropathy will be evaluated. It evaluates 8 items: inflammation and duration of this, pain, muscle atrophy and strength, crackles, and loss of flexion and extension. It has a score of 0 (no joint damage) to 20 points (maximum joint damage) per joint (elbows, knees and ankles). A gait rating is added to the 120 points (range 0-4 points), the maximum rating on this scale being 124 points
Change from baseline functionality after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With the Timed Up and Go Test, basic mobility skills, strength, balance and agility will be evaluated. This test can help predict an individual's risk of falls and other adverse outcomes. This test measures the time it takes for a patient to get up from a chair (without using their arms to get up), walk to a line on the floor 3 m away, turn around, and return to the chair and sit down. Two measurements will be made per patient and the best value will be used for analysis. The unit of measurement is seconds, where the shorter the time, the better the score.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No